CLINICAL TRIAL: NCT04729907
Title: A Long-Term Extension Study of Nusinersen (BIIB058) Administered at Higher Doses in Participants With Spinal Muscular Atrophy Who Previously Participated in an Investigational Study With Nusinersen
Brief Title: A Study to Learn About the Long-Term Safety of Higher Doses of Nusinersen (BIIB058) Given as Injections to Participants With Spinal Muscular Atrophy (SMA) Who Took Part in an Earlier Nusinersen Trial (ONWARD)
Acronym: ONWARD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 232SM302; 2023-505637-27 (Other: EU CTIS)
Expanded Access: NCT02865109 (No longer available)
Record Dates: First submitted 2020-12-11; First posted 2021-01-29 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIIB058 28 mg (Prior Maintenance Dose 28 mg) (Experimental): Participants who received maintenance dose of 28 milligrams (mg) nusinersen in study 232SM203 (NCT04089566), will receive maintenance dose of 28 mg nusinersen, by intrathecal injection, on Day 1, followed by maintenance dose of 28 mg nusinersen, by intrathecal injection, every 4 months, up to Day 1921.
  Interventions: Drug: Nusinersen
- BIIB058 50/28 mg (Prior Maintenance Dose 12 mg) (Experimental): Participants who received maintenance dose of 12 mg nusinersen in study 232SM203 (NCT04089566), will receive loading dose of 50 mg nusinersen, by intrathecal injection, on Day 1, followed by maintenance dose of 28 mg nusinersen, by intrathecal injection, every 4 months, up to Day 1921.
  Interventions: Drug: Nusinersen

INTERVENTIONS:
Drug: Nusinersen — Administered as specified in the treatment arm
  Other Names: BIIB058; Spinraza

SUMMARY:
In this study, researchers will learn more about the use of nusinersen (BIIB058) in participants with spinal muscular atrophy (SMA). This study is an extension study and will enroll only those participants who have completed treatment in the parent study, 232SM203.

The main goal of the study is to learn about the long-term safety of nusinersen. The main questions researchers want to answer are:

* How many participants have adverse events and serious adverse events during the study?
* How do the results of electrocardiograms (ECGs), vital signs, and laboratory tests including blood and urine tests change after treatment?
* How many participants have a low platelet count after treatment?
* How many participants had a change in the time it took for their heart to recharge between beats after treatment?
* How does each participant's height and other measures of growth change after treatment?
* How much do the results of neurological exams that check movement, reflexes, and brain function change after treatment?

Researchers will also learn about the effect of nusinersen on mobility using various tests. They will study body movements, reflexes, balance, and coordination. They will also record if participants need help with breathing.

The 232SM302 study will be done as follows:

* Participants will be screened to check if they can join the study.
* Participants will receive their 1st dose of nusinersen in this study about 4 months after their final dose in the parent study.
* Each participant will receive nusinersen once every 4 months during the treatment period.
* Nusinersen will be given through a lumbar puncture, which involves injecting the drug into the fluid around the spinal cord in the lower back.
* The treatment period will last for up to 64 months (1921 days).
* There will be a follow-up safety period that lasts from 4 to 8 weeks.
* In total, participants will have up to 19 study visits. Participants will stay in the study for close to 6 years.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the long-term safety and tolerability of nusinersen administered intrathecally at higher doses to participants with spinal muscular atrophy (SMA) who previously participated in study 232SM203 (NCT04089566).

The secondary objective of this study is to evaluate the long-term efficacy of nusinersen administered intrathecally at higher doses to participants with SMA who previously participated in study 232SM203 (NCT04089566).

ELIGIBILITY:
Key Inclusion Criteria:

* Completed the Day 302 visit in study 232SM203 (NCT04089566) in accordance with the study protocol

Key Exclusion Criteria:

* Treatment with another investigational therapy or enrollment in another interventional clinical study
* Treatment with an approved therapy for SMA after the Day 302 Visit of Study 232SM203 (NCT04089566)

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 1921
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a birth defect, or is a medically important event.
Change from Baseline in Growth Parameters | Up to Day 1921
  Growth parameters will be assessed by measuring body length or height (if feasible and appropriate), ulnar length (all participants), and head circumference, chest circumference, and arm circumference (all participants 3 years of age and younger) in centimeters.
Number of Participants With Shifts from Baseline in Clinical Laboratory Parameters | Up to Day 1921
Number of Participants With Shifts from Baseline in Electrocardiogram (ECG) | Up to Day 1921
Number of Participants With Shifts from Baseline in Vital Signs | Up to Day 1921
Change from Baseline in Activated Partial Thromboplastin Time (aPTT) | Up to Day 1921
Change from Baseline in Prothrombin Time (PT) | Up to Day 1921
Change from Baseline in International Normalized Ratio (INR) | Up to Day 1921
Change from Baseline in Urine Total Protein | Up to Day 1921
Change from Baseline in Neurological Examination Outcomes for Participants ≤2 Years of Age | Up to Day 1921
  For participants 2 years of age and younger, the Hammersmith Infant Neurological Exam (HINE) Sections 1 and 3 will be conducted. This standard examination (developed by [Dubowitz and Dubowitz 1981]) is a quantitative scorable method for assessing the neurological development of infants between 2 and 24 months of age. The examination includes assessment of cranial nerve functions, posture, movements, tone, and reflexes. The HINE Section 1 form utilized in ONWARD contains 26 items and the Section 3 form utilized contains 3 items. For HINE Section 1 items, each item is scored 0-3. For HINE Section 3 items, scoring is variable (1-4, 1-5, or 1-6). Higher scores indicate better neurological function.
Number of Participants with Change from Baseline in Neurological Examination Outcomes for Participants >2 Years of Age | Up to Day 1921
  For all participants >2 years of age, standard neurological examinations, which include assessments of mental status, level of consciousness, sensory function, motor function, cranial nerve function, and reflexes, will be conducted.
Percentage of Participants With a Postbaseline Platelet Count Below the Lower Limit of Normal on at least 2 Consecutive Measurements | Up to Day 1921
Percentage of Participants With a Postbaseline Corrected QT Interval Using Fridericia's Formula (QTcF) of >500 millisecond (msec) and an Increase from Baseline to Any Postbaseline Timepoint in QTcF of >60 msec | Up toDay 1921

SECONDARY OUTCOMES:
Total Number of New World Health Organization (WHO) Motor Milestones | Up to Day 1921
Number of Participants Who Used Respiratory Support, by Type | Up to Day 1921
Number of Hours Per Day of Respiratory Support | Up to Day 1921
Number of Days That Respiratory Support Is Used | Up to Day 1921
Time to Death (Overall Survival) | Up to Day 1921
Change from Baseline in Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) Total Score | Up to Day 1921
  The CHOP INTEND test is designed to evaluate the motor skills of infants with significant motor weakness. It includes 16 items (capturing neck, trunk, and proximal and distal limb strength) structured to move from easiest to hardest with the grading including gravity eliminated (lower scores) to antigravity movements (higher scores). All item scores range from 0-4. The total score ranges from 0-64, with higher scores depicting better response. This outcome measure will be assessed for participants who were evaluated with this measure in study 232SM203 (NCT04089566).
Change from Baseline in Hammersmith Infant Neurological Examination (HINE) Section 2 Motor Milestones | Up to Day 1921
  Section 2 of the HINE is used to assess motor milestones of the participants. It is composed of 8 motor milestone categories: voluntary grasp (0 to 3), ability to kick in supine position (0 to 4), head control (0 to 2), rolling (0 to 3), sitting (0 to 4), crawling (0 to 4), standing (0 to 3), and walking (0 to 3). Total HINE score is the sum of points from each item and can range from 0 to 26, with higher scores depicting better level of ability. This outcome measure will be assessed for participants who were evaluated with this measure in study 232SM203 (NCT04089566).
Percentage of HINE Section 2 Motor Milestone Responders | Up to Day 1921
  Section 2 of HINE is used to assess motor milestones of participants. It is composed of 8 motor milestone categories: voluntary grasp (0 to 3), ability to kick in supine position (0 to 4), head control (0 to 2), rolling (0 to 3), sitting (0 to 4), crawling (0 to 4), standing (0 to 3), and walking (0 to 3). Total HINE score is sum of points from each item and can range from 0 to 26, with higher scores depicting better level of ability. HINE section 2 motor milestone responder is participant who demonstrates at least 2-point increase in category of ability to kick or increase to maximal score on that category or 1-point increase in motor milestones category of head control, rolling, sitting, crawling, standing, or walking, and among 7 motor milestone categories (excluding voluntary grasp), participant demonstrates improvement in more categories than worsening. This outcome measure will be assessed for participants who were evaluated with this measure in study 232SM203 (NCT04089566).
Percentage of Time Spent on Ventilation | Up to Day 1921
  This outcome measure will be assessed for participants who were evaluated with this measure in study 232SM203 (NCT04089566).
Time to Death or Permanent Ventilation | Up to Day 1921
  Permanent ventilation is defined as tracheostomy or ≥16 hours of ventilation/day continuously for >21 days in the absence of an acute reversible event. This outcome measure will be assessed for participants who were evaluated with this measure in study 232SM203 (NCT04089566).
Change from Baseline in Hammersmith Functional Motor Scale - Expanded (HFMSE) Score | Up to Day 1921
  The HFMSE is a tool used to assess motor function in children with SMA. The original 20 item Hammersmith Functional Motor Scale (HFMS) was expanded to include 13 additional items to improve sensitivity for the higher functioning ambulant population. Participants will be asked to complete a specific movement and are then graded on the quality and execution of that movement. Higher scores indicate higher levels of motor ability. The overall score is the sum of the scores for all activities, with a maximum score of 66 with higher scores depicting better ability to perform activities. Participants ≥ 2 years of age (at the time of the study visit) will be evaluated with HFMSE.
Change from Baseline in Revised Upper Limb Module (RULM) Score | Up to Day 1921
  The RULM is developed to assess upper limb functional abilities participants with SMA. This test consists of upper limb performance items that are reflective of activities of daily living. The RULM is scored from 0 to 37 points, with higher scores indicating better function. Participants ≥ 2 years of age (at the time of the study visit) will be evaluated with RULM.
Change From Baseline in Plasma Levels of Neurofilament (NF) | Up to Day 1921

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (39):
- United States (7):
  - Stanford University Medical Center, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Medical Center, Plano, Texas
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital das Clinicas - FMUSP, São Paulo
- London Health Sciences Centre (LHSC) - Children's Hospital, London, Ontario, Canada
- Chile (3):
  - Hospital Luis Calvo Mackenna, Santiago
  - Clinica Las Condes, Santiago
  - Clinica MEDS La Dehesa, Santiago
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Guangzhou Woman and Children's Medical Center, Guangzhou, Guangdong
  - The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Hospital Universitario San Ignacio, Bogotá, Colombia
- Tallinn Children's Hospital, Tallinn, Estonia
- Germany (2):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen, Hesse
- Italy (2):
  - Fondazione Serena Onlus - Centro Clinico Nemo, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Japan (3):
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Hyogo Medical University Hospital, Nishinomiya-shi, Hyōgo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo-To
- Saint George University Hospital Medical Center, Beirut, Lebanon
- Mexico (3):
  - Instituto Nacional de Pediatria, Mexico City, Mexico City
  - Hospital Infantil de Mexico Federico Gomez, Mexico City, Mexico City
  - Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
- Russia (2):
  - Russian Children Neuromuscular Center of Veltischev, Moskva
  - Regional Pediatric Clinical Hospital #1, Yekaterinburg
- Saudi Arabia (3):
  - King Fahad Specialist Hospital, Dammam
  - National Guard Health Affairs: King Abdulaziz Medical City, Jeddah
  - King Faisal Specialist Hospital & Research Center, Riyadh
- Spain (3):
  - Hospital Sant Joan de Deu, Esplugues Del Llobregat, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- See also: SMA Europe — https://www.sma-europe.eu/
- See also: CureSMA — https://www.curesma.org/
- See also: Muscular Dystrophy Association — http://www.mda.org/disease/spinal-muscular-atrophy